CLINICAL TRIAL: NCT03022591
Title: Management of Twins With Short Cervix at a Single Institution: A Retrospective Review
Brief Title: Short Cervix - Twins
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Laura Vricella, MD, Principal investigator, St. Louis University
Other Study IDs: 27027
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Short Cervix
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Management — management of twin pregnancies with a short cervix diagnosed between 16 0/7 WGA to 27 6/7 WGA.

SUMMARY:
This is a retrospective chart review. The purpose of this study will be to look at the outcomes of twin pregnancies diagnosed with short cervix along with the intervention (treatment) that these patients received.

DETAILED DESCRIPTION:
In 2010, the incidence of preterm birth in twin gestations was 23% before 34 weeks and 58% before 37 weeks, while the overall incidence of PTB in all pregnancies was only 3.41% and 11.5%, respectively. Twin gestations are also at increased risk of being low birth weight infants.

Goldenberg et al demonstrated in 1996 that a cervical length less than 25 mm at 24 weeks gestation in twin pregnancies was the best predictor of preterm birth at <32 weeks, <35 weeks, and < 37 weeks. In 1999, Souka et al reported that in twin pregnancies with a cervical length less than 15 mm at 23 weeks gestation, the preterm birth rate <32 weeks was approximately 66%.

A Cochrane Review from 2014 concluded that placing a cerclage is not associated with a significant difference regarding perinatal deaths or neonatal morbidity, but this analysis was for all forms of cerclage in multiple gestations (physical examination-indicated, history-indicated, and ultrasound-indicated). It did also state "ultrasound-indicated cerclage appears to be associated with an increased risk for the composite adverse neonatal outcome, including respiratory distress syndrome, low and very low birthweight, given there is no evidence of a consistent subgroup effect, the observed results can most likely be attributed to chance."

In a 2015 retrospective cohort study of twin pregnancies with asymptomatic short cervix, Amanda Roman et al demonstrate similar results to those of the Cochrane Review for patients with CL <25 mm. However, they did show a trend towards prolonged pregnancy, decreased spontaneous PTB <34 weeks, and fewer NICU admissions for a subset of patients with CL < 15 mm that received a cerclage compared to control.

In February 2016, Goya et al investigated the role of the pessary for women with twin gestations and short cervix diagnosed via ultrasound. A significant reduction in the rate of preterm birth prior to 34 weeks was found in the pessary group (16.2% vs 39.4%), with no significant differences in neonatal morbidity or mortality.

Chart review will collect information documented on the data collection sheet, including medical and OB history, current pregnancy course, treatment for short cervix and information on hospitalization including labor and delivery, postpartum course and neonatal birth information.

The investigators will analyses and compare this group of women using short cervix diagnosis, management decisions and outcomes during the antepartum period, labor, delivery and post partum course for possible signs and symptoms of those at risk for Pre Term Birth and outcomes of their infants.

ELIGIBILITY:
Inclusion Criteria:

* Charts of all women who had twins and a short cervix will be reviewed,

Exclusion Criteria:

* singleton

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 14-55yrs of age Female all ethnic backgrounds
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Short cervix | 1 year
  management decisions and outcomes of twin pregnancies diagnosed with short cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Laure Vricella, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No